CLINICAL TRIAL: NCT06536127
Title: Prospective Monocentric Study Evaluating the Circulating NK Cells Phenotype and the ImmunoScore® in Patients With Non Metastatic Rectal Adenocarcinoma Treated With Preoperative Radiochemotherapy With or Without Initial Chemotherapy
Brief Title: Prospective Monocentric Study Evaluating the Circulating NK Cells Phenotype and the ImmunoScore® in Patients With Non Metastatic Rectal Cancer
Acronym: IMMUNOREC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Sainte Catherine (Other)
Responsible Party: Principal Investigator, Recherche clinique, Principal Investigator, Institut Sainte Catherine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ICAP
Record Dates: First submitted 2024-07-29; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Rectal Cancer; Non Metastatic Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Blood samples
  Interventions: Diagnostic Test: Blood samples

INTERVENTIONS:
Diagnostic Test: Blood samples — Nk cells and ImmunoScore

SUMMARY:
Until 2020, the standard treatment for rectal cancer was a combination of radiotherapy and concomitant chemotherapy based on IV or oral 5FU, with a low complete response rate.

The randomised phase 3 PRODIGE 23 trial evaluated a regimen of FOLFIRINOX chemotherapy prior to neoadjuvant RTCT, with 3-year disease-free survival as the primary endpoint. Patients in the PRODIGE 23 arm had significantly better 3-year disease-free survival (76% versus 69%; p=0.034) and 3-year metastasis-free survival (79% versus 72%; p=0.017) than patients in the standard arm, and the complete histological response rate to neoadjuvant treatment (ypT0N0) doubled from 12% in the standard arm to 28% in the PRODIGE 23 arm.

The main benefit of surgical de-escalation is to improve patients' quality of life. The main obstacle to the non-surgical management of these patients with a complete response after RTCT was the impact on survival in the event of local recurrence. Habr-Gama et al. showed that the WW strategy, combined with close follow-up, resulted in excellent disease control in the event of local recurrence, with organ conservation in almost 80% of patients.

The selection of patients eligible for this non-surgical treatment (Wait and Watch WW) remains the main issue, which is why some physicians are still reluctant to adopt it.

The immune cells known to be involved in the anti-tumour response are T lymphocytes, B lymphocytes and Natural Killers (NK). These cells play a crucial role in the initiation, development and progression of cancers. They are naturally considered as potential targets for immunotherapy, but also as biological markers.

In several tumour types, particularly colorectal cancers, it has been shown that a CD8+ lymphocyte infiltrate in the tumour is associated with a better prognosis. NK cells have also been studied in the circulating blood of colorectal cancer patients and have been shown to be predictive of 3-year survival. These results suggest that prognosis may depend more on the quality of the anti-tumour immune response than on clinical parameters.

The prognosis of adenocarcinoma of the rectum is essentially estimated by TNM uicc staging. It needs to be better estimated in order to adapt treatments to the risk of relapse. The beneficial effect of the immune response developed by the patient against colorectal tumours is certainly an important area of research.

The INSERM U1183 unit is developing a technology for analysing blood NK cells and their phenotype, including those acquired by trogocytosis (WO/2016/005548). The aim of our study will be to compare the phenotype of circulating NK cells in patients with rectal cancer before, during and after treatment, and to study the relationship with relapse-free survival and the rate of complete clinical response in non-operated patients and histological response in operated patients.

A clinically applicable immunological test called 'Immunoscore®' quantifies the density of two types of immune cells in the tumour and its invasion front: total T lymphocytes (CD3+) and killer lymphocytes (cytotoxic CD8+). The aim of the international study published in The Lancet was to assess the prognostic value of the Immunoscore test in patients with colon cancer. Given the major performance of this test in colorectal cancer, researchers are currently evaluating the Immunoscore test in rectal cancer and studying its ability to predict response to neoadjuvant treatment in rectal cancer. El sissy et al. reported very encouraging results on the predictive value of the test for rectal tumours in complete response after radio-chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years

Histologically proven adenocarcinoma of the rectum

Patient with rectal cancer (cT2-4N0 or cT1-T4N+)

Patients whose planned treatment is: standardised CTRT comprising 50Gy intensity-modulated irradiation and Capecitabine with or without additional dose (contact therapy). Neoadjuvant chemotherapy with FOLFOX or FOLFIRINOX may be given prior to RTCT.

IMRT-type radiotherapy treatment

Women of childbearing age must provide proof of effective contraception (sterilisation for you and/or your partner, transdermal, vaginal, oral, subcutaneous or injectable hormonal contraception and intrauterine devices).

Person affiliated to or benefiting from a social security scheme.

Free, informed and written consent signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research).

Exclusion criteria:

Metastatic disease

Unresectable disease

History of pelvic irradiation or contraindication to pelvic irradiation

Contraindications to the administration of one of the following chemotherapy drugs: irinotecan, oxaliplatin, or 5 FU, capecitabine

Presence of an evolving concomitant neoplasia other than the following: i/ treated in situ cervical cancer, ii/ spino or basal cell skin cancer, iii/ cancer in complete remission for more than 3 years.

Psychological, social, family or geographical conditions preventing compliance with the study protocol and follow-up examinations.

Persons under legal protection (guardianship, curatorship, safeguard of justice)

Persons deprived of their liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between clinical and survival data and tests results | 5 years

SECONDARY OUTCOMES:
Nk cells kinetics evaluation during course of treatment | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- ICAP, Avignon, France

IPD SHARING:
Plan to Share IPD: No